CLINICAL TRIAL: NCT00313547
Title: Impact of High-Dose Quinapril Versus Low-Dose Quinapril Plus Amlodipine on Autonomic Regulation and on Sympathetic Activation in Response to Cold Exposure in Hypertensive Patients With Impaired Glucose Tolerance, Diabetes or Coronary Artery Disease
Brief Title: High-Dose Quinapril Versus Low-Dose Quinapril Plus Amlodipine in the Treatment of High-Risk Hypertensive Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Very difficult to recruit patients/slow recruitment(2 patients in nearly 2 years).
Sponsor: Montreal Heart Institute (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MHI 05740; Pfizer NRA9060008; (Investigator initiated study)
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2007-08

CONDITIONS: Hypertension
Keywords: Blood pressure; Hypertension; Renin; Aldosterone; Heart rate variability
MeSH Terms: conditions — Hypertension | interventions — Quinapril; Amlodipine

INTERVENTIONS:
Drug: Quinapril 40 mg
Drug: Quinapril 10 mg and amlodipine 5 mg

SUMMARY:
The purpose of this study is to compare the impact of two blood pressure lowering treatments (high dose quinapril versus low dose quinapril plus amlodipine) on variations in heart rate over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented history of hypertension defined as: SBP > or = 140 mmHg or DBP > or = 90 mmHg if hypertension untreated or patients currently treated for hypertension.
* Documented CAD or diabetes or impaired glucose tolerance
* Sinus rhythm

Principal Exclusion Criteria:

* Previous intolerance or allergic reaction to an ACE inhibitor, an ARB or dihydropyridine calcium channel blocker
* History of angioedema or cough related to previous ACE inhibitor use.
* Systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg in untreated patients
* Systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg in patients currently treated by an ACE inhibitor or an ARB
* Creatinine clearance < 30 ml/min
* Significant liver dysfunction
* Current serum potassium > or = 5 mmol/L or a history of marked ACE inhibitor or ARB induced hyperkalemia resulting in either a serum potassium > or = 5.5 mmol/L or a life-threatening adverse event.
* History of HF or known LVEF < or = 45%
* Bilateral renal artery stenosis (or unilateral if only one kidney)
* Unstable angina, myocardial infarction or coronary revascularization within the last 3 months.
* Connective tissue disease or chronic inflammatory condition
* Active malignancy
* Active infection in the last 2 weeks
* Inability or any contraindication to perform an exercise test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Heart rate variability

SECONDARY OUTCOMES:
Tolerability
Renin, aldosterone
MMPs
Oxidative stress
Norepinephrine
Lactate
Exercise tolerance at 20 and -8 degree celsius
Blood pressure
Impact of selected pharmacogenetic polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Michel White, MD, Principal Investigator — Montreal Heart Institute; Simon de Denus, B. Pharm, MSc, Principal Investigator — Faculty of Pharmacy, University of Montreal/Montreal Heart Institute; Jacques de Champlain, MD, PhD, Principal Investigator — Faculty of Medicine, University of Montreal
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada